CLINICAL TRIAL: NCT02700048
Title: Intra-nasal Naloxone for Treatment of Impaired Awareness of Hypoglycemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: research grant for the trial was not funded
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1103M96932
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Hypoglycemia Unawareness; Type 1 Diabetes
Keywords: type 1 diabetes; hypoglycemia; hypoglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 3 doses of intra-nasal saline will be given during controlled hypoglycemic insulin clamps
  Interventions: Drug: Intra-nasal saline
- Treatment with intra-nasal Naloxone (Experimental): 3 doses of intra-nasal naloxone (4 mg each) will be given during controlled hypoglycemic insulin clamps
  Interventions: Drug: intra-nasal naloxone

INTERVENTIONS:
Drug: intra-nasal naloxone — 3 doses of intra-nasal naloxone (4 mg each) will be given during controlled hypoglycemic insulin clamps
  Other Names: Narcan
  Arms: Treatment with intra-nasal Naloxone
Drug: Intra-nasal saline — 3 doses of intra-nasal saline will be given during controlled hypoglycemic insulin clamps
  Arms: Placebo

SUMMARY:
This is a single center, single-blind randomized cross over design trial that will compare the impact of intra-nasal naloxone vs. intra-nasal saline administration during experimental hypoglycemia on day one on responses to experimental hypoglycemia on day two. Investigators intend to enroll 18 individuals to obtain the complete data sets from 15 participants. Expected duration of subject participation is 10-12 weeks. This study will consist of two 2-day intervention visits separated by approximately 8 weeks.

DETAILED DESCRIPTION:
This is a single center, single-blinded randomized cross over design trial, that will compare the impact of IN naloxone vs. IN saline during experimental hypoglycemia on day one on the responses to experimental hypoglycemia on day two. 18 participants will be studied twice, 8 weeks apart. On each occasion participants will undergo a 2 hour hypoglycemic clamp (target 50 mg/dl) in the morning and in the afternoon on day one and then again on the morning of day 2. During the morning clamps, samples will be collected for later measurement of serum epinephrine, glucagon and cortisol levels and participants will be asked to complete a hypoglycemia symptom questionnaire. 3 intranasal doses (4 mg each) of naloxone hydrochloride or IN saline will be administered to the subject on day 1. Plasma will be collected for measurement of naloxone concentrations on day 1 primary outcome is the difference in peak epinephrine secretion during the morning episodes of hypoglycemia on days one and two, thus each participant will have two observations: one from their naloxone experiment and one from their saline experiment.

Secondary endpoint will be naloxone pharmacokinetics including maximum concentration (Cmax), time to maximum concentration (Tmax) and area under the curve (AUC)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are capable of giving informed consent.
2. Female subjects must be post-menopausal for at least 1 year, or surgically incapable of bearing children, or practicing at least one or more of the following methods of contraception for three months prior to, and during the study: hormonal, intrauterine device (IUD), or barrier method in combination with a spermicide.
3. Subject should be medication free, other than hormonal birth control, for 48 hours before through 24 hours after study drug administration. If the need for medication is identified during this time period, it will be discussed with and approved by the PI.

Exclusion Criteria:

1. Women who are pregnant.
2. Women who are breastfeeding.
3. Subject has a known hypersensitivity to naloxone.
4. Subject with hypertension
5. Subject has a significant history of cardiac, neurologic, psychiatric, oncologic, endocrine, metabolic, renal or hepatic disease
6. Subject has taken or used any investigational drug or device in the 30 days prior to screening.
7. Subject has taken either prescribed or over the counter medication for 48 hours prior to study drug administration on either of the study days, other than hormonal birth control.
8. History of narcotic or heroin abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moheet, MD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants consented, but only 3 actually started the trial
Period: Overall Study
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3
Not completed — The device failed so the study wasn't completed and participants were dropped | 0 | 3

BASELINE CHARACTERISTICS:
Population: the device failed so data was not collected and participants dropped prior to collecting baseline data
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Within Person Difference in Peak Epinephrine During Hypoglycemia
Description: Primary endpoint will be the within person difference in peak epinephrine secretion during the morning episodes of hypoglycemia on days one and two; investigators will compare this difference between the two treatment conditions
Time Frame: 2 years
Population: the device failed so data was not collected and participants dropped
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Naloxone Pharmacokinetics
Description: maximum concentration (Cmax)
Time Frame: 2 year
Population: the device failed so data was not collected and participants dropped
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Naloxone Pharmacokinetics
Description: area under the curve (AUC)
Time Frame: 2 year
Population: the device failed so data was not collected and participants dropped
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: the device failed so data was not collected and participants dropped
Description: the device failed so data was not collected and participants dropped
Arm/Group | Placebo | Treatment With Intra-nasal Naloxone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02700048/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT02700048/ICF_001.pdf